CLINICAL TRIAL: NCT00301782
Title: Randomized Phase II Trial of Intensive Induction Chemotherapy (CBOP/BEP) and Standard BEP Chemotherapy in Poor Prognosis Male Germ Cell Tumors
Brief Title: Combination Chemotherapy in Treating Male Patients With Germ Cell Tumors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medical Research Council (Other Government)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000456203; MRC-TE23; EU-205107; ISRCTN53643604; EUDRACT-2004-000405-22
Record Dates: First submitted 2006-03-09; First posted 2006-03-13 (Estimated); Last update posted 2013-08-26 (Estimated); Status verified 2007-05

CONDITIONS: Extragonadal Germ Cell Tumor; Teratoma; Testicular Germ Cell Tumor
Keywords: testicular choriocarcinoma and embryonal carcinoma; testicular choriocarcinoma and teratoma; testicular choriocarcinoma and yolk sac tumor; testicular choriocarcinoma; testicular embryonal carcinoma and teratoma; testicular embryonal carcinoma and yolk sac tumor; testicular embryonal carcinoma; testicular yolk sac tumor; testicular yolk sac tumor and teratoma; stage I malignant testicular germ cell tumor; stage II malignant testicular germ cell tumor; stage III malignant testicular germ cell tumor; recurrent malignant testicular germ cell tumor; recurrent extragonadal non-seminomatous germ cell tumor; stage I extragonadal non-seminomatous germ cell tumor; stage II extragonadal non-seminomatous germ cell tumor; stage III extragonadal non-seminomatous germ cell tumor; stage IV extragonadal non-seminomatous germ cell tumor; recurrent extragonadal germ cell tumor; testicular immature teratoma; testicular mature teratoma; adult teratoma
MeSH Terms: conditions — Teratoma; Testicular Germ Cell Tumor; Carcinoma, Embryonal; Endodermal Sinus Tumor; Testicular Neoplasms | interventions — Bleomycin; Carboplatin; Cisplatin; etoposide phosphate; Vincristine

INTERVENTIONS:
Biological: bleomycin sulfate
Drug: carboplatin
Drug: cisplatin
Drug: etoposide phosphate
Drug: vincristine sulfate

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as cisplatin, vincristine, bleomycin, carboplatin, and etoposide phosphate, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving more than one drug (combination chemotherapy) may kill more tumor cells. It is not yet known which combination chemotherapy regimen is more effective in treating germ cell tumors.

PURPOSE: This randomized phase II trial is studying two different combination chemotherapy regimens to compare how well they work in treating male patients with germ cell tumors.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare the response rate in patients with poor-prognosis extracranial nonseminoma germ cell tumors treated with intensive induction chemotherapy comprising cisplatin, vincristine, bleomycin, and carboplatin followed by bleomycin, etoposide phosphate, and cisplatin (BEP) vs standard BEP chemotherapy.

Secondary

* Compare overall and progression-free survival of patients treated with these regimens.
* Compare the toxicity of these regimens in these patients.

OUTLINE: This is a multicenter, open-label, randomized study. Patients are stratified according to participating center, pre-protocol low-dose chemotherapy (yes vs no), and other clinically important factors. Patients are randomized to 1 of 2 treatment arms.

* Arm I (BEP): Patients receive bleomycin IV over 15 minutes once on day 1 or 2 and days 8 and 15 and etoposide phosphate IV over 1 hour and cisplatin IV over 4 hours on days 1-5. Treatment repeats every 21 days for up to 4 courses in the absence of disease progression or unacceptable toxicity.
* Arm II (CBOP/BEP): Patients receive chemotherapy according to the following schedule:

  * Weeks 1-6: Patients receive cisplatin IV over 6 hours on days 1, 2, 8, 15, 16, and 22 (OR over 4 hours on days 1-5 and 15-19); vincristine IV on days 1, 8, 15, 22, 29, and 36; bleomycin IV over 15 minutes on days 1, 15, 29, and 36 and bleomycin IV continuously on days 8-12 and 22-25; and carboplatin IV over 30-60 minutes on days 8 and 22.
  * Weeks 7-15: Patients receive bleomycin IV continuously on days 1-5, 8-12, and 15-19 and etoposide phosphate IV over 1 hour and cisplatin IV over 4 hours on days 1-5. Treatment repeats every 21 days for 4 courses.

After completion of study treatment, patients are followed periodically for 5 years.

Peer Reviewed and Funded or Endorsed by Cancer Research UK

PROJECTED ACCRUAL: A total of 88 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Nonseminoma germ cell tumor of any extracranial primary site diagnosed by 1 of the following methods:

  * Histologic confirmation
  * Alpha-fetoprotein (AFP) > 1,000 ng/mL or human chorionic gonadotropin (hCG) > 5,000 IU/L with appropriate clinical picture in a man < 45 years of age
* Poor prognosis features as defined by ≥ 1 of the following:

  * AFP > 10,000 ng/mL
  * hCG > 50,000 IU/L
  * Lactic dehydrogenase > 10 times normal
  * Nonpulmonary visceral metastases
  * Mediastinal primary site

PATIENT CHARACTERISTICS:

* Male
* WHO performance status 0-3
* Glomerular filtration rate > 50 mL/min

  * Less than 50 mL/min eligible if due to obstructive neuropathy that can be relieved by stenting or nephrostomy
* No comorbid condition that would prevent treatment
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

* No prior chemotherapy except low-dose chemotherapy to stabilize disease before study therapy

Min Age: 16 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2005-06; Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Response rates to treatment

SECONDARY OUTCOMES:
Overall survival
Progression-free survival
Toxicity

CONTACTS AND LOCATIONS:
Overall Officials: Robert A. Huddart, MD, Study Chair — Royal Marsden NHS Foundation Trust
Locations (20):
- United Kingdom (20):
  - Queen Elizabeth Hospital at University Hospital of Birmingham NHS Trust, Birmingham, England
  - Bristol Haematology and Oncology Centre, Bristol, England
  - Addenbrooke's Hospital, Cambridge, England
  - Gloucestershire Oncology Centre at Cheltenham General Hospital, Cheltenham, England
  - Walsgrave Hospital, Coventry, England
  - Royal Devon and Exeter Hospital, Exeter, England
  - Leeds Cancer Centre at St. James's University Hospital, Leeds, England
  - Leicester Royal Infirmary, Leicester, England
  - Saint Bartholomew's Hospital, London, England
  - University College of London Hospitals, London, England
  - Christie Hospital, Manchester, England
  - Clatterbridge Centre for Oncology, Merseyside, England
  - Nottingham City Hospital, Nottingham, England
  - Rosemere Cancer Centre at Royal Preston Hospital, Preston, England
  - Berkshire Cancer Centre at Royal Berkshire Hospital, Reading, England
  - Southampton General Hospital, Southampton, England
  - Royal Marsden - Surrey, Sutton, England
  - Beatson West of Scotland Cancer Centre, Glasgow, Scotland
  - Raigmore Hospital, Inverness, Scotland
  - Velindre Cancer Center at Velindre Hospital, Cardiff, Wales

REFERENCES:
- [Result] Huddart RA, Gabe R, Cafferty F, et al.: A randomized phase II trial of intensive induction chemotherapy (CBOP/BEP) and standard BEP in poor prognosis germ cell tumors (MRC TE23, CRUK 05/014, ISRCTN53643604). [Abstract] J Clin Oncol 29 (Suppl 15): A-4508, 2011.